CLINICAL TRIAL: NCT00264628
Title: An Outpatient, Randomised, Double-blind, Placebo Controlled, Parallel Group Exploratory Study to Evaluate Safety, Tolerability and Efficacy of GW679769 in Patients With Fibromyalgia Syndrome Comorbid With Depression.
Brief Title: GW679769 In Fibromyalgia
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: SND103929
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Depressive Disorder; Depression; Fibromyalgia
Keywords: NK1-antagonist; Depression; Fibromyalgia; GW679769; Outpatient
MeSH Terms: conditions — Depressive Disorder; Depression; Fibromyalgia | interventions — casopitant

INTERVENTIONS:
Drug: GW679769

SUMMARY:
The purpose of the study is to investigate safety, tolerability and efficacy of oral GW679769 up to 120 mg dose compared to placebo in patients with ACR(American College of Rheumatology)-defined fibromyalgia, co-morbid with depression.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of fibromyalgia (ACR criteria).
* Non-severe depression (HAM-D score >14 <24).
* Women must commit to consistent use of an acceptable method of birth control.

Exclusion criteria:

* Severe depression (HAM-D score > 24).
* Unable to discontinue medications for pain or depression.
* Laboratory and ECG value at screening outside sponsor defined ranges.
* Positive to stool occult blood test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire (FIQ) total score | throughout study

SECONDARY OUTCOMES:
Effect of GW679769 vs placebo in health-related quality of life outcomes | throughout study
Relationship between PK of GW679769 and clinical outcome in patients | throughout study
Safety and Tolerability | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline